CLINICAL TRIAL: NCT04351035
Title: Retrospective, Multi-center Cross-sectional Study on Paediatric Central Nervous Systerm Tumours by CNOG-MC001 Collaborative Group
Brief Title: National Wide Cross-sectional Study in Paediatric Central Nervous System Tumours in China -- the CNOG-MC001 Registry
Status: Completed | Type: Observational
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: CNOG-MC001 Collaborative Group (Unknown)
Responsible Party: Principal Investigator, Jie Ma, MD, PhD, Director of Dept Pediatric Neurosurgery, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: CNOG-MC001
Record Dates: First submitted 2020-04-16; First posted 2020-04-17 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Tumors, Central Nervous System; Pediatric Brain Tumor; Malignant Brain Tumor; Benign Brain Tumor
Keywords: national wide; cross-sectional; retrospective; CNOG-MC001; pediatric; central nervous system tumor
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with CNS tumours: Patients newly diagnosed with CNS tumours in children younger than 18 y/o, who were under in-patient treatment, were labeled as candidate cases in the CNOG-MC001 cohort for reviewing.
  Interventions: Procedure: Tumour resection

INTERVENTIONS:
Procedure: Tumour resection — It is mandatory that patients recieve surgical treatment for pathological diagnosis of CNS tumours in enrolled patients. Surgical resection of tumours could be regarded as total / subtotal / partial resection and biopsy.

SUMMARY:
Tumours of central nervous system (CNS) is the most common type of solid tumour in childhood. In China, there is limited epidemiology information. Released data from Chinese CDC did not include types of CNS tumours and geographic contribution. As the Children's Neuro-Oncology Group (CNOG) was established in China in May 2017, it makes studies from multiple centers in children's brain tumors become practical. This retrospective cross-sectional study was aligned on CNOG annual meeting in 2018 and research group was named as CNOG-MC001 (MC, multicenter) collaborative group.

DETAILED DESCRIPTION:
CNS tumours are mostly seen solid tumours in childhood , as the second common malignancy following leukemia in children. The annual age-standardized incidence rate per 1,000,000 person-years (ASR) of CNS tumour in international children's cancer incidence study is 20-30. In Asia, ASR of paediatric CNS tumours is around 15.0-24.9 in Japan, Korea, Singapore. For Chinese races including mainland of China, Taiwan and Hong Kong, ASRs of paediatric CNS tumour are 15.0, 17.4 and 23.8.

In 2017 in Shanghai, Children's Neuro-Oncology Group (CNOG) was found in 5th CSPN (Chinese Society of Pediatric Neurosurgery) / 9th CPNF (China Pediatric Neurosurgery Forum) conference, with 35 founding member institutions and 30 founding observation member institutions in mainland of China. Based on this progress, national wide registry (CNOG-MC001) was settled to obtain basic information about CNS tumour cases, combined with available epidemiology data from publications to assess current medical situation on paediatric CNS tumours in China. The protocol of CNOG-MC001 was aligned by CSPN and CNOG member institutions in CNOG annual meeting in 2018 and the study ofiicially started right after the meeting on 20181027.

The first step of this study is a national wide pre-survey to all 35 CNOG member institutions and other 22 CSPN members. The pre-survey data sheet included number of annual surgically treated paediatric CNS tumour cases (age ranging from 0 to 18 years old, classified by WHO Classification of Tumours of the Central Nervous System 2016 version), to assess the proper sites to be involved in this study. After retrieving the pre-survey results, large-scale, detailed case data sheets will be sent to participating institutions as members of CNOG-MC001 collaborative group.

ELIGIBILITY:
Inclusion Criteria:

* patients who were newly diagnosed with CNS tumour admitted for in-patient treatments during period of Jan.1st 2016 to Dec. 31st 2017
* patients who were less than 18 year-old at diagnosis
* patients with available mandatory information as age, gender during enrollment
* patients must have pathological diagnosis of tumours, which followed 2016 edition of the World Health Organization (WHO) Classification of Tumours of the Central Nervous System (CNS), except the following conditions:

  1. Diffuse Intrinsic Pontine Glioma (DIPG) according to classic symptoms and typical MRI
  2. confirmed NF1 patients with classic symtoms and MRI representing Optic Pathway Glioma (OPG) with no surgical treatment indications will be marked as "pilocytic astrocytoma"
  3. patients with newly diagnosed recurrence or metastasis of previously confirmed (before Jan.1st 2016) Embryonal Tumours (medulloblastoma, emryonal tumour with multilayered rosettes - C19MC altered, atypical teratoid / rhabdoid tumour / others) and high grade gliomas (glioblastoma, anaplastic astrocytoma) that were unwilling to recieve second surgical treatment / inoperable / without surgical indication, will be marked as original diagnosis
  4. patients with newly diagnosed relapse of previously confirmed (before Jan.1st 2016) low grade glioma (defined as pilocytic astrocytoma, diffuse astrocytoma, pilomyxoid astrocytoma, pleomorphic xanthoastrocytoma, subependymal giant cell astrocytoma, oligodendroglioma, oligoastrocytoma, ganglioglioma, desmoplastic infantile astrocytoma and ganglioglioma, dysembryoplastic neuroepithelial tumour, papillary glioneuronal tumour, rosette-forming glioneuronal tumour of the fourth ventricle, angiocentric glioma, dysplastic cerebellar gangliocytoma, extraventricular neurocytoma, cerebellar liponeurocytoma, and central neurocytoma) and ependymal tumours in cross-sectional period, who were unwilling to be operated / inoperable / without surgical indication, will be marked as original diagnosis
* clinical, image and pathology data of patients with unidentified pathological diagnosis from member sites of CNOG-MC001 collaborative group will be sent to study center for reviewing; cases with unidentifiable diagnosis after center review and alignment with CNOG-MC001 sites will be marked as "unknown"

Exclusion Criteria:

* confirmed CNS metatasis patients whose tumour tissues were obtained from other systems other than CNS will be excluded
* patients with newly diagnosed recurrence or metastasis of previously confirmed CNS Tumours, will be excluded when primary tumour diagnosis and progression time points were both in cross-sectional period; these patients will be only enrolled as "newly diagnosed cases with primary tumours" and recorded as "progressed in follow-up" in follow-up data sheet
* patients with newly diagnosed relapse of previously confirmed (before Jan.1st 2016) low grade glioma and ependymal tumours, who were unwilling to be operated / inoperable, and were suspected as malignant transformation, will be excluded due to lack of pathological diagnosis
* patients with insufficient or inconsistant data (e.g: patient diagnosed with primary medulloblastoma with tumour located in cerebral) will be excluded in center review after consulting with data-upload institutions

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Newly diagnosed paediatric (0-18 y/o) CNS tumous in period of Jan.1st 2016 to Dec.31st 2017, with sufficient baseline data and clear pathological diagnosis according to classification of CNS tumours - WHO 2016 version (for exceptions please refer to eligibility criteria)
Sampling Method: Non-Probability Sample
Enrollment: 4303 (Actual)
Dates: Start 2018-10-27 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Baseline information of children with CNS tumours | 2 years
  Baseline information including gender, age, and institutional geographic data are required for epidemiology analysis.
Tumour type and anatomic location | 2 year
  Tumour type according to 2016 edition of the World Health Organization (WHO) Classification of Tumours of the Central Nervous System (CNS) is mandatory for epidemiology analysis.

SECONDARY OUTCOMES:
Overall Survival | 1 year
  Available overall survival data with post surgery treatments records of enrolled cases is preferred but not mandatory for outcome analysis.
Progression Free Survival | 1 year
  Progression free survival data is preferred but not mandatory for outcome analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Jie MA, M.D., Ph.D., Study Chair — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (38):
- China (38):
  - Anhui Provincial Children's Hospital, Hefei, Anhui
  - Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - the First Hospital Affiliated To Army Medical University, Chongqing, Chongqing Municipality
  - Army Medical Center of PLA, Chongqing, Chongqing Municipality
  - the First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - 900 Hospital of the Joint Logistics Team of PLA, Fuzhou, Fujian
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - Guangdong 999 Brain Hospital, Guangzhou, Guangdong
  - Affiliated Hospital of Guilin Medical University, Guilin, Guangxi
  - Affiliated Hospital of Zunyi Medical College, Zunyi, Guizhou
  - the Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - the First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Children's Hospital Affiliated to Zhengzhou University, Zhengzhou, Henan
  - the Third Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science & Technology, Wuhan, Hubei
  - Renmin Hospital of Wuhan University / Hubei General Hospital, Wuhan, Hubei
  - the Fifth Affiliated Hospital of Zhengzhou University, Zhengzhou, Hunan
  - the Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - the First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Jiangxi Provincial Children's Hospital, Nanchang, Jiangxi
  - the First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - the First Bethune Hospital of Jilin University, Ch’ang-ch’un, Jilin
  - Shengjing Hospital Affiliated to China Medical University, Shenyang, Liaoning
  - the General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Xi'an Children's Hospital, Xi'an, Shaanxi
  - Xijing Hospital of Air Force Military Medical University, Xi'an, Shaanxi
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Qilu Children's Hospital of Shandong University, Jinan, Shandong
  - Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Xinhua Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Children's Hospital of Fudan University, Shanghai, Shanghai Municipality
  - the Children's Hospital of Shanxi Province, Taiyuan, Shanxi
  - Sichuan Academy of Medical Sciences & Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan
  - People's Hospital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang Uygur Autonomous Region
  - Kunming Children's Hospital, Kunming, Yunnan
  - the Children's Hospital, Zhejiang University School of Medicine, Hanzhou, Zhejiang